CLINICAL TRIAL: NCT04510155
Title: Liver Glycogen Dynamics and Substrate Oxidation in Lean Healthy Volunteers
Brief Title: Liver Glycogen Dynamics
Acronym: LGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Charlotte Andriessen, Principal Investigator, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL72118.068.20
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Glycogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short overnight fast (Experimental): Overnight fasting duration intervention: Participants will receive their last evening meal at 11 pm and stay overnight fasted afterwards for (9.5h).
  Interventions: Behavioral: Overnight fasting duration
- Long overnight fast (Experimental): Overnight fasting duration intervention: Participants will receive their last evening meal at 4.30 pm and stay overnight fasted afterwards for (16h).
  Interventions: Behavioral: Overnight fasting duration

INTERVENTIONS:
Behavioral: Overnight fasting duration — Subjects will adhere to overnight fasting protocol for 1 day

SUMMARY:
The purpose of this study is to investigate the effect of prolonged overnight fasting in the hepatic glycogen stores

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Caucasian (people will be excluded when having a ≥50% racial African/Asian background)
* Participants should have suitable veins for cannulation or repeated venipuncture
* Women are post-menopausal (defined as at least 1 year post cessation of menses)
* Men and women aged ≥ 45 and ≤ 75 years at the start of the study
* Body mass index (BMI) 18.5 - 25 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months)
* Sedentary lifestyle (not more than 3 hours of vigorous sports per week)

Exclusion Criteria:

* Type 2 Diabetes Mellitus
* Active diseases (cardiovascular, diabetes, liver, kidney, cancer or other)
* Any contraindication for MRI scanning
* Alcohol consumption of >2 servings per day
* Regular smoking
* No use of medication interfering with investigated study parameters (as determined by responsible physician)
* Participants who do not want to be informed about unexpected medical findings, or do not wish that their physician

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Hepatic glycogen content | 1 hour
  Measured with 13C-MRS

SECONDARY OUTCOMES:
Substrate oxidation | 14 hours
  Measured as RQ

OTHER OUTCOMES:
Intrahepatic fat content and composition (1H-MRS) | 30 minutes
  Measured with 1H-MRS
De novo lipogenesis (DNL) | 20 hours
  measured as percentage of palmitate in VLDL-TG originating from DNL
Hepatic fat oxidation | 5 hours
  measured as plasma BHB levels
Liver volume | 5 minutes
  Measured with MRI
Substrate oxidation | 30 minutes
  measured with indirect calorimetry
Plasma metabolites related to energy metabolism | 5 hours
  measured in plasma samples
Body composition | 5 minutes
  fat mass/fat free mass measured with BodPod

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, Dr, Principal Investigator — Principal Investigator
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No